CLINICAL TRIAL: NCT04011137
Title: The Effect of Upper-body High-intensity Interval Training on Postprandial Metabolic Control in Persons With Chronic Paraplegia
Brief Title: High-intensity Interval Training and Mixed Meal Responses in Persons With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Bilzon, Professor, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EP 17/18 141
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Paraplegia
Keywords: high-intensity interval training; postprandial metabolism
MeSH Terms: conditions — Paraplegia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No exercise - 30-min of rest
- High-intensity interval training (Experimental): 8 x 60 s intervals at 70% peak power output (intersperesed with 60 s recovery intervals at 10% peak power output)
  Interventions: Other: Exercise
- Moderate-intensity continous training (Experimental): 25 min at 45% peak power output
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Arm-cranking exercise
  Arms: High-intensity interval training; Moderate-intensity continous training

SUMMARY:
Persons with chronic paraplegia at an increased risk of developing cardiovascular disease and type-2 diabetes compared to the able-bodied population. There is mounting evidence from the able-bodied literature that high-intensity interval training (HIIT) is more effective than moderate-intensity continuous training (MICT) at improving markers of cardiometabolic health. Before we can understand the long-term training effects of HIIT in this population, it is important to compare the acute metabolic responses to a typical mixed-macronutrient meal following both exercise modalities.

This study is recruiting adults (aged 18-65 years) with paraplegia (T2 or below) who sustained their spinal cord injury more than one-year ago. Participants will need to attend the laboratory at the University of Bath on four separate occasions, once for preliminary testing, and three times for study trials.

DETAILED DESCRIPTION:
The aim of this research is to determine the metabolic responses to a mixed-meal tolerance test following a bout of HIIT and MICT in persons with chronic paraplegia. The hypothesis is that HIIT and MICT will be more effective at reducing the total triglyceride responses compared to a resting control condition.

Preliminary measurements:

Preliminary testing will include anthropometric measurements of supine length, weight, waist and hip circumferences, and resting blood pressure. There will also be an assessment of resting metabolic rate, sub-maximal and maximal exercise capacity, and a HIIT familiarisation session. All of the exercise protocols will take place on an arm crank ergometer at the University of Bath.

Physical activity monitoring:

For 7 days, participants will be fitted with a physical activity monitor (Actiheart™). Participants should not make any conscious changes to their normal lifestyle habits/routines during this period.

Main trial days:

In the 2 days prior to the main trial day, participants will be asked to record their food and drink intake and 48 hours before they should refrain from performing any strenuous physical activity. In the 24 hours prior participants should also refrain from consuming any alcohol or caffeine.

Following a 10-hour overnight fast, an expired gas sample and venepuncture blood sample will be taken prior to exercise. Participants will then perform a bout of HIIT, MICT or a resting control condition. Following exercise, a cannula will be inserted into a vein and baseline blood sample(s) taken for analysis of metabolic markers.

The participant will then be asked to consume a smoothie, consisting of peanut butter, banana, coconut oil, sugar, and chocolate-flavoured whey protein powder. The meal should be consumed within 10 minutes and blood samples will be taken from the cannula at 15, 30, 45 60, and 90 minutes and then at every hour for 6 hours after consumption of the meal to monitor changes in metabolic and inflammatory markers. Expired gas samples will also be taken hourly and indirect calorimetry will be used to estimate relative fat and carbohydrate metabolism in response to the meal.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a chronic (>12 months post-injury) SCI below T2
* Individuals who spend >75% of their waking day in a wheelchair
* Weight stable (weight not changed by >3% over the last 3 months)

Exclusion Criteria:

* Individuals who an acute (<12 months post-injury) SCI
* Individuals who spend <75% of their waking day in a wheelchair
* Individuals on type-2 diabetes medication
* Individuals with a peanut allergy
* Individuals who self-report use of lipid-lowering agents
* Individuals self-reporting active medical issues (pressure sores, urinary tract infections, cardiac disorders, musculoskeletal complaints of the upper extremities, or cardiovascular contraindications to exercise testing)
* Individuals who report uncontrolled or regular autonomic dysreflexia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Postprandial triglyceride concentrations | 6 hours
  Postprandial triglyceride concentrations in serum samples

SECONDARY OUTCOMES:
Postprandial glucose concentrations | 6 hours
  Postprandial glucose concentrations in serum samples
Postprandial insulin concentrations | 6 hours
  Postprandial insulin concentrations in serum samples
Postprandial non-esterified fatty acid concentrations | 6 hours
  Postprandial non-esterified fatty acid concentrations in serum samples
Postprandial substrate oxidation | 6 hours
  Postprandial substrate oxidation determined by indirect calorimetry
Rating of Perceived Exertion | MICT: End of Warm-Up, 6 minutes 15 seconds, 12 minutes 30 seconds, 18 minutes 45 seconds, End of Exercise. HIIT: End of Warm-Up, 8 minutes, 12 minutes, 16 minutes, 20 minutes)
  Global, central, and local rating of perceived exertion during exercise
Heart Rate | MICT: End of Warm-Up, 6 minutes 15 seconds, 12 minutes 30 seconds, 18 minutes 45 seconds, End of Exercise. HIIT: End of Warm-Up, 8 minutes, 12 minutes, 16 minutes, 20 minutes)
  Heart rate during exercise
Affect | MICT: End of Warm-Up, 6 minutes 15 seconds, 12 minutes 30 seconds, 18 minutes 45 seconds, End of Exercise. HIIT: End of Warm-Up, 8 minutes, 12 minutes, 16 minutes, 20 minutes)
  Affect measured through the Feeling Scale (FS) during exercise. FS is a one item scale ranging from +5 ("Very good") to -5 ("Very bad").
Exercise Enjoyment | 30 minutes post-exercise
  Enjoyment measured by the Physical Activity Enjoyment Scale (PACES). PACES is a 17-item scale, with each item scored from 1 to 7. The total score will be calculated.
Self-efficacy | 30-minutes post-exercise
  Confidence in ability to perform exercise performed during trial in the next 4 weeks measured using a 5-item scale ranging from 0% ("Not at all" to 100% ("Extremely confident").

CONTACTS AND LOCATIONS:
Overall Officials: James Bizon, Principal Investigator — University of Bath
Locations (1):
- Department for Health, Bath, United Kingdom

REFERENCES:
- [Derived] Farrow MT, Maher JL, Nightingale TE, Thompson D, Bilzon JLJ. A Single Bout of Upper-Body Exercise Has No Effect on Postprandial Metabolism in Persons with Chronic Paraplegia. Med Sci Sports Exerc. 2021 May 1;53(5):1041-1049. doi: 10.1249/MSS.0000000000002561. PMID 33560775